CLINICAL TRIAL: NCT02428127
Title: Efficacy of a Carbohydrate Drink on Speed, Agility and Power in School Going Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 203093
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Growth and Development
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): 20g Carbohydrate powder fortified with multiple micronutrients, reconstituted as a beverage in 200mL lukewarm water. This will be administered twice a day
  Interventions: Dietary Supplement: Carbohydrate beverage powder
- Calorie matched protein powder (Active Comparator): 20g Calorie matched protein powder with 80% protein, reconstituted as a beverage in 200mL lukewarm water. This will be administered twice a day
  Interventions: Dietary Supplement: Calorie matched beverage powder
- Control (Placebo Comparator): 200mL lukewarm water given twice a day
  Interventions: Other: Water

INTERVENTIONS:
Dietary Supplement: Carbohydrate beverage powder — Carbohydrate beverage powder fortified with multiple micronutrients. 20g of study product will be administered orally twice a day
  Arms: Test
Dietary Supplement: Calorie matched beverage powder — Calorie matched beverage powder with 80% protein.20g of study product will be administered orally twice a day
  Arms: Calorie matched protein powder
Other: Water — lukewarm water
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the impact of a beverage containing carbohydrate powder fortified with micronutrients on agility, speed, and power in school going children

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by participant's parents or legally accepted representative
* Good general health
* Non anemic children (Hb≥12 g/dl)
* Academy/development level athlete (at least 3 activity sessions per week, for a minimum of 2 hours of activity in each session e.g. hockey, football, team sports)

Exclusion Criteria:

* Child in care
* Allergy/Intolerance to study materials
* History of cardiovascular disorder, respiratory diseases, diabetes mellitus, serious infection/injuries/surgeries (within past 3 months)
* Participation in any nutritional study in past 1 year
* Substance abuse
* Children on any kind of medication in past 1 month of screening

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Agility fatigue index | Baseline and 4h post-baseline
  Agility fatigue index (FI) will be calculated from Repeat Agility Performance Test, using 'Brower equipment'. This assessment includes a 24 meter agility run, repeated on 6 occasions, with every sprint and recovery interval lasting for 65 seconds (eg. if the first agility effort takes the participant 5 seconds, they will have 55 seconds to return to start line for a 5 seconds countdown before their second agility effort). Agility FI=[100X(total agility time÷ideal agility time)]-100. Here, ideal agility time is the best agility time for each participant multiplied by number of repetitions

SECONDARY OUTCOMES:
Change from baseline in Speed fatigue index | Baseline and 4h post-baseline
  Speed fatigue index (FI) will be calculated from Repeat Sprint Performance Test, using 'Brower equipment'. This assessment includes a 30 meter sprint, repeated on 6 occasions, with every sprint and recovery interval lasting for 65 seconds (eg. if the first sprint takes the participant 5 seconds, they will have 55 seconds to return to start line for a 5 second countdown before their second sprint). Speed FI=[100X(total speed time÷ideal speed time)]-100. Here, ideal speed time is the best speed time for each participant multiplied by number of repetitions
Change from baseline in Mean power output | Baseline and 4h post-baseline
  Mean power output (MPO) will be calculated from Wingate Anaerobic Test, using 'Cycle ergometer'. The participant is allowed to pedal at a constant pace, without resistance and then with additional weights (resistance). This is repeated on three occasions. Overall MPO=(sum of MPO from 3 repetitions at baseline)-(sum of MPO from 3 repetitions at post treatment).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Pune, India

REFERENCES:
- [Background] http://www.i-scholar.in/index.php/Ijnd/article/view/130266